CLINICAL TRIAL: NCT01777360
Title: Bicentric Prospective Study, Evaluating Bronchial THERMOPLASTY in a Patient Presenting Severe Uncontrolled Asthma
Acronym: ASMATHERM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P 120102
Record Dates: First submitted 2013-01-17; First posted 2013-01-28 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Asthma
Keywords: severe; uncontrolled
MeSH Terms: conditions — Asthma; Lymphoma, Follicular | interventions — Bronchial Thermoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- THERMOPLASTY (Experimental): ALAIR, radiofrequency catheter for bronchial THERMOPLASTY
  Interventions: Device: ALAIR, radiofrequency catheter for bronchial THERMOPLASTY

INTERVENTIONS:
Device: ALAIR, radiofrequency catheter for bronchial THERMOPLASTY — radiofrequency catheter for bronchial THERMOPLASTY

SUMMARY:
To determine, from patients presenting severe asthma and an increase in bronchial smooth muscle mass, those who would be the best candidates for bronchial THERMOPLASTY. THERMOPLASTY should improve control of the asthma, reduce day-to-day symptoms and severe exacerbations, and improve respiratory function

DETAILED DESCRIPTION:
Bicentric prospective study, evaluating bronchial THERMOPLASTY in patients with severe uncontrolled asthma and significant bronchial smooth muscle mass. Primary Objective is to determine patients who would be the best candidates for bronchial THERMOPLASTY which should improve control of the asthma, reduce day-to-day symptoms and severe exacerbations, and improve respiratory function. Primary Endpoint will be the reduction in smooth muscle surface area, objectified on bronchial biopsies before and after THERMOPLASTY in patients presenting severe asthma and secondary criteria are:

* number of severe exacerbations (with oral corticosteroids, emergency room visits, hospitalizations)
* time until the first exacerbation
* respiratory function
* control of the asthma (ACQ - Asthma Control Questionnaire)
* quality of life (AQLQ - Asthma Quality of Life Questionnaire)
* fraction of exhaled nitric oxide (FENO)
* measurement of the thickness of the bronchial wall using tomodensitometry (scan). The inclusion of period of 28 months is limited to a maximum of 80 subjects. The actual number will be determined using the two-stage stop method. An intermediate analysis will be carried out following the evaluation and statistical analysis of the 40 patients.
* If the primary endpoint p-value is <0.0294, success will be declared and the inclusions will cease.
* If the p-value is >0.0294, additional patients will be recruited up to a total of 80 patients included and assessed. At inclusion, sociodemographic data will be collected, number of exacerbations per year, date of fibroscopy, data on asthma control (ACQ), data on quality of life (AQLQ), respiratory function (EFR), fraction of exhaled nitric oxide (FENO), thickness of the bronchial wall evaluated using scanner and surface area of smooth muscle in the bronchial sub-mucous layer will be evaluated. At 3 months post-THERMOPLASTY, same data will be collected. One year after THERMOPLASTY, number of exacerbations, data on asthma control (ACQ),and quality of life (AQLQ), respiratory function (EFR), fraction of exhaled nitric oxide (FENO), thickness of the bronchial wall and possible complications will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* Patients with severe asthma that is uncontrolled despite optimal treatment and who have presented at least one exacerbation while taking oral corticosteroids within the previous 12 months
* With a variable bronchial obstruction (FEV1 >30 and <70% of theoretical)
* Patients known to have severe asthma under the care of the Pneumology Department of BICHAT Hospital in Paris (Prof. AUBIER) and the Nord Hospital in Marseilles (Prof. CHANEZ).
* Covered by French national health insurance.

Exclusion Criteria:

* Patient having had severe exacerbation of their asthma requiring high doses of oral corticosteroids (> 60 mg) during the month before inclusion.
* Patient with exacerbation.
* Patient having presented a severe exacerbation or other undesirable reactions related to a bronchoscopy.
* Patient having an FEV1 <30% of theoretical after taking a short-acting B2 mimetic. - Patient having oxygen saturation measured by pulse oximetry <90% in ambient air.
* Patient presenting clinically significant electrocardiogram abnormalities.
* Patient presenting an uncontrolled co-morbidity.
* Patient presenting coagulation and platelet abnormalities.
* Patient having a habitual contraindication to a bronchial endoscopy.
* Patient having hemostasis disorders
* Presence of a pacemaker, internal defibrillator, or other implantable electronic device.
* Contraindication to corticosteroids at high doses and atarax
* Pregnant women and lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
smooth muscle surface area | 3 month after THERMOPLASTY
  Reduction in smooth muscle surface area, objectified on bronchial biopsies before and after THERMOPLASTY in patients presenting severe asthma.

SECONDARY OUTCOMES:
respiratory function | 12 month after thermoplasty
  number of severe exacerbations

CONTACTS AND LOCATIONS:
Overall Officials: Aubier Michel, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Bichat Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Debray MP, Dombret MC, Pretolani M, Thabut G, Alavoine L, Brillet PY, Taille C, Khalil A, Chanez P, Aubier M. Early computed tomography modifications following bronchial thermoplasty in patients with severe asthma. Eur Respir J. 2017 Mar 15;49(3):1601565. doi: 10.1183/13993003.01565-2016. Print 2017 Mar. PMID 28298402